CLINICAL TRIAL: NCT06096168
Title: Ambispective Study Evaluating the Clinical Results of SAGITTA EVL R Revision Stems
Acronym: 2022-10
Status: Completed | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-10_Sagitta EVL-R
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: Hip Arthropathy
Keywords: Total Hip Prosthesis Revision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This clinical study is conducted to collect data on hip arthroplasty with the SAGITTA EVL-R revision femoral stems manufactured by SERF. In order to reflect current practice, a comprehensive and continuous series of patients will be included.

This study will confirm the performance and safety of the SAGITTA EVL R revision femoral stems within the framework of MDR 2017/745 and in relation to the recommendations of the MEDDEV guide 2.7.1. Rev 4 (Clinical Evaluation Guide), which provides for a systematic procedure to monitor clinical data in order to verify the claimed performance of medical devices.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old at the time of surgery,
* Patient implanted with a SAGITTA EVL R revision femoral stem within its indications between 01/01/2016 and 31/12/2018,
* Affiliated to French health insurance system

Exclusion Criteria:

* Patient who has not expressed consent for data collection and participation in the study,
* Patient unable to understand the surgeon's instructions or to perform postoperative follow-up.
* Patient with a contraindication to the use of the SAGITTA EVL R revision femoral stem
* Patient implanted with a SAGITTA EVL R revision femoral stem outside its indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects who needed a revision of total hip arthroplasty, implanted with a SAGITTA EVL-R revision femoral stem according to instructions for use, over a period of time between 31/01/2016 and 31/12/2018.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Rouen - Hôpital Charles Nicolle, Rouen, Seine Maritime, France

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: 42
Groups:
- Per Protocol Population: All patients implanted with a SAGITTA EVLR revision stem in CHU Rouen between 2016 and 2018 meeting inclusion/exclusion criteria. All patients are included in the same arm. No randomization, no control arm.
Period: Overall Study
Arm/Group | Per Protocol Population
Started | 42; 42 42 (Number of unit is corresponding to : Operated Hips)
Completed | 10; 10 42 (Number of unit is corresponding to : Operated Hips)
Not Completed | 32; 32 42
Not completed — Death | 30
Not completed — Revision | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: number of implants
Groups:
- Per Protocol Population: All patients implanted with a SAGITTA EVLR revision stem in CHU Rouen between 2016 and 2018 meeting inclusion/exclusion criteria
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 42
Number analyzed (number of implants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.4 (8.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Weight [Mean (Standard Deviation); unit: kg] — Population: Weight not available for 3 patients (3 hips)
  kg
    number analyzed (Participants) | 39
    (all) | 72.8 (19.0)

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate at Mid Term Follow-up
Description: Assess the survival rate, at least 4 year-follow-up, whatever the cause of revision. Cumulative survival rate expressed in percentage of implants not revised (remaining in place) using Kaplan Meier calculation.
Time Frame: Between 4 to 7 years after surgery
Measure: Number; unit: percentage of implant survival
Units Other Than Participants: number of implants
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 42
Number analyzed (number of implants) | 42
percentage of implant survival | 90.1

2. Secondary Outcome: Adverse Events
Description: List type and frequency of complications, investigated by clinical and radiological examination following investigator's usual practice
Time Frame: From per operative period to 4/6 years after surgery
Measure: Number; unit: participants
Units Other Than Participants: hips implanted
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 42
Number analyzed (hips implanted) | 42
participants
  Sepsis | 1
  Greater trochanter fracture | 1
  Posterior dislocation - vicious attitude of the hip | 1
  Femoral fracture | 1
  Fracture with greater trochanter displacement | 1

3. Secondary Outcome: Survival Rates at Mid Term Follow-up (by Component)
Description: Assess the survival rates at least, 4 year-follow-up, whatever the cause of revision, regarding each component of the prothesis
Time Frame: At 4/6 years after surgery
Measure: Number; unit: percentage of implant survival
Units Other Than Participants: number of hips
Groups:
- Per Protocol Population Implanted With NOVAE COPTOS Femoral Cup: All patients implanted with a SAGITTA EVLR revision stem in CHU Rouen between 2016 and 2018 meeting inclusion/exclusion criteria and with NOVAE COPTOS femoral cup
Arm/Group | Per Protocol Population Implanted With NOVAE COPTOS Femoral Cup
Number analyzed (Participants) | 7
Number analyzed (number of hips) | 7
percentage of implant survival | 100

4. Secondary Outcome: Survival Rates at Mid Term Follow-up (by Etiology)
Description: Assess the survival rates at least, 4 year-follow-up, whatever the cause of revision, regarding etiology.
  Percentage of patients with implant in place dispatched following reason for implantation
Time Frame: At 4/6 years after surgery
Measure: Number; unit: percentage of implant
Units Other Than Participants: hips implanted
Groups:
- Population Concerned by Revision + Osteosynthesis With Wires: All patients implanted with a SAGITTA EVLR revision stem in CHU Rouen between 2016 and 2018 meeting inclusion/exclusion criteria concerned by Revision + osteosynthesis with wires
Arm/Group | Population Concerned by Revision + Osteosynthesis With Wires
Number analyzed (Participants) | 5
Number analyzed (hips implanted) | 5
percentage of implant | 80

5. Secondary Outcome: Patient's Satisfaction
Description: Assessed by the surgeon through questionary with a 5 item-scale : very satisfied / satisfied / neither satisfied - nor unsatisfied / unsatisfied / very unsatisfied
Time Frame: At 4/6 years after surgery
Measure: Number; unit: number of hips
Units Other Than Participants: hips implanted
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 10
Number analyzed (hips implanted) | 10
number of hips
  Very satisfied | 4
  Rather satisfied | 4
  Neither satisfied nor unsatisfied | 2
  Rather unsatisfied | 0
  Very unsatisfied | 0

6. Secondary Outcome: Oblivion of Prosthesis
Description: Assess the degree of forgetfulness of the prosthesis using FJS-score (Forgotten Joint Score) :
  FJS stands for Forgotten Joint Score. The Forgotten Joint Score assessment consists of 12 questions and is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities
Time Frame: At 4/6 years after surgery
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: hips implanted
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 9
Number analyzed (hips implanted) | 9
score on a scale | 80.4 (10.15)

7. Secondary Outcome: Functional Improvement
Description: Evaluate pain, walking, limping and activities of daily life using Harris Hip Score :
  The global Harris Hip Score consists of a 0 to 100 points scale (100 points is the better outcome)
Time Frame: At 4/6 years after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hips implanted
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 9
Number analyzed (hips implanted) | 9
score on a scale | 71.5 (21.45)

ADVERSE EVENTS:
Time Frame: Until >4-years follow up (maximum duration of 90 months)
Arm/Group | Per Protocol Population
All-Cause Mortality (participants affected / at risk) | 30/42
Serious Adverse Events (participants affected / at risk) | 4/42
Other Adverse Events (participants affected / at risk) | 1/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Per Protocol Population (N=42)
Sepsis (Infections and infestations) | 1 (1)
Posterior dislocation (Surgical and medical procedures) | 1 (1)
Femoral fracture (Surgical and medical procedures) | 1 (1)
Fracture with greater trochanter displacement (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Per Protocol Population (N=42)
Greater trochanter fracture (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT06096168/Prot_000.pdf